CLINICAL TRIAL: NCT04132141
Title: Effect of Immersive Virtual Reality Breaks on Shift-worker Alertness
Brief Title: VR Breaks on Shift-worker Alertness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Neal Sikka, Associate Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 051818
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Each recruited subject completes 6 shifts with observation. Half the shifts have normal or wild type breaks, the other half are virtual reality breaks. The order is random.
Masking Description: all data is collected by the Research assistant and de-identified. The investigator will not know which data belongs to which participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR intervention (Other): each subject will be own control. subjects breaks will be randomly assigned to VR or WT until they complete 3 for each type or a total of 6
  Interventions: Other: Virtual Reality Headset with curated content

INTERVENTIONS:
Other: Virtual Reality Headset with curated content — clinicians will wear VR immersive headset for up to 15 minutes during their break

SUMMARY:
Physician wellness is a hot topic today. Fatigue and alertness are common challenges faced during long work hours. Virtual reality is an immersive technology which has been demonstrated to distract people from pain, stress, and anxiety. Guided relaxation and meditation can impact alertness. There is no literature reporting the impact immersive technologies like VR sessions could have on alertness, a critical area of concern in health care today which impacts physician wellness, quality of care, and duty hours.

The investigator's long-term goal is to develop solutions that can be used across industries to improve human alertness. To solve this problem, the investigators propose to test the feasibility of using an immersive virtual reality experience as a scheduled break and measure the interventions effect on post-break alertness, stress, and anxiety. Previous work at our Institution has demonstrated that VR experiences can reduce pain, stress and anxiety in patients presenting to the emergency department.

DETAILED DESCRIPTION:
Physician wellness is a hot topic today. Fatigue and alertness are common challenges faced during long work hours. Virtual reality is an immersive technology which has been demonstrated to distract people from pain, stress, and anxiety. Guided relaxation and meditation can impact alertness. There is no literature reporting the impact immersive technologies like VR sessions could have on alertness, a critical area of concern in health care today which impacts physician wellness, quality of care, and duty hours.

The investigator's long-term goal is to develop solutions that can be used across industries to improve human alertness. To solve this problem, the investigator proposes to test the feasibility of using an immersive virtual reality experience as a scheduled break and measure the interventions effect on post-break alertness, stress, and anxiety. Previous work at our Institution has demonstrated that VR experiences can reduce pain, stress and anxiety in patients presenting to the emergency department.

Hypothesis: Short immersive VR breaks are expected to increase alertness and reduce stress and anxiety in residents, physicians, and medical students working on shifts as compared to unstructured breaks.

Aim 1 will establish a biometric footprint of activities relating to the shift of a resident, physician, medical student, or nurse. Understanding how biometric parameters change when performing different activities will establish a baseline for comparing the effect of immersive VR breaks.

Aim 2 will seek to tag the activities a resident, physician, medical student, or nurse is performing during the shift to add context to the biometric data

Aim 3 will be to evaluate metrics for alertness, stress and anxiety of a resident, physician, medical student, or nurse during their shift and specifically determine how they change with immersive VR intervention

The proposed study will establish a new model for managing physician alertness, stress and anxiety and provide insights into viable and effective interventions to improve these parameters for other occupations. The expected improvement in alertness and reduction in stress and anxiety could be highly impactful in creating a safer workplace. These methods will also help derive biometric maps of physician activities that could be used for a variety of physician wellness interventions. The impact of this study could be wide reaching in occupational health.

ELIGIBILITY:
Inclusion Criteria:

* GW residents, physicians, medical students, and nurses between the ages of 18-65.
* will have at least 5 shifts over the study period in the GW Hospital

Exclusion Criteria:

* Unable to consent to study due to cognitive difficulty
* Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware and software
* Sensitivity to flashing light or motion
* Pregnancy, or a medical condition where the participant is prone to frequent nausea or dizziness
* Recent stroke
* Injury to the eyes, face, neck, or arms that prevents comfortable use of VR hardware or software, or safe use of the hardware (e.g., open sores, wounds, or skin rash on face)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Psycho-motor Vigilance Testing (PVT) | PVT will be collected in each study shift and compared at the end of the study period about 4 months
  response time measure of alertness using PVT software

SECONDARY OUTCOMES:
Alertness | Alertness will be collected in each study shift and compared at the end of the study period about 4 months
  Self Reported level of alertness using 10 point Likert scale
Stress | Stress will be collected in each study shift and compared at the end of the study period about 4 months
  Self Reported level of stress using 10 point Likert scale
Anxiety | Anxiety will be collected in each study shift and compared at the end of the study period about 4 months
  Self Reported level of anxiety using 10 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Neal K Sikka, MD, Principal Investigator — George Washington University
Locations (1):
- GW Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith-Coggins R, Howard SK, Mac DT, Wang C, Kwan S, Rosekind MR, Sowb Y, Balise R, Levis J, Gaba DM. Improving alertness and performance in emergency department physicians and nurses: the use of planned naps. Ann Emerg Med. 2006 Nov;48(5):596-604, 604.e1-3. doi: 10.1016/j.annemergmed.2006.02.005. Epub 2006 May 2. PMID 17052562
- [Background] Alhola P, Polo-Kantola P. Sleep deprivation: Impact on cognitive performance. Neuropsychiatr Dis Treat. 2007;3(5):553-67. PMID 19300585
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Han T, Nag A, Simorangkir RBVB, Afsarimanesh N, Liu H, Mukhopadhyay SC, Xu Y, Zhadobov M, Sauleau R. Multifunctional Flexible Sensor Based on Laser-Induced Graphene. Sensors (Basel). 2019 Aug 9;19(16):3477. doi: 10.3390/s19163477. PMID 31395810
- [Background] Langelotz C, Scharfenberg M, Haase O, Schwenk W. Stress and heart rate variability in surgeons during a 24-hour shift. Arch Surg. 2008 Aug;143(8):751-5. doi: 10.1001/archsurg.143.8.751. PMID 18711034